CLINICAL TRIAL: NCT00838799
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study of the Safety and Efficacy of RGH-896 in Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: Study of the Safety and Efficacy of RGH-896 in Patients With Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: James Perhach, Ph.D., Executive Director, Clinical Development, Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG8-MD-02
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: diabetic; peripheral; neuropathic; pain; chronic; diabetes
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome; Diabetes Mellitus | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: RGH-896
- 2 (Experimental)
  Interventions: Drug: RGH-896
- 3 (Experimental)
  Interventions: Drug: RGH-896
- 4 (Active Comparator)
  Interventions: Drug: pregabalin
- 5 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RGH-896 — 45 mg TID, capsules, 14 weeks.
  Arms: 1
Drug: RGH-896 — 30 mg TID, capsules, 14 weeks.
  Arms: 2
Drug: RGH-896 — 15 mg TID, capsules, 14 weeks.
  Arms: 3
Drug: pregabalin — 100 mg, TID, capsules, 14 weeks.
  Other Names: Lyrica
  Arms: 4
Drug: placebo — TID, capsules, 14 weeks.
  Arms: 5

SUMMARY:
This study is designed to evaluate the safety and efficacy of RGH-896 in patients with diabetic peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 to 75 years of age
* A diagnosis of painful diabetic neuropathy
* Controlled blood glucose
* Willingness to wash out all analgesic medications used for DPNP
* Female patients either postmenopausal, surgically sterile, or practicing a medically acceptable method of contraception
* Female patients who are not pregnant

Exclusion Criteria:

* Acute infections or cardiac problems
* Past use of pregabalin
* History of severe psychiatric disorder
* History of any amputation due to diabetes
* History of seizure disorder
* Active diabetic foot ulcers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in mean daily pain rating | Baseline to Week 14

SECONDARY OUTCOMES:
50% reduction in pain | Baseline to Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Gage, PhD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Locations (54):
- United States (54):
  - Forest Investigative Site, Birmingham, Alabama
  - Forest Investigative Site, Mesa, Arizona
  - Forest Investigative Site, Tempe, Arizona
  - Forest Investigative Site, Jonesboro, Arkansas
  - Forest Investigative Site, Little Rock, Arkansas
  - Forest Investigative Site, North Little Rock, Arkansas
  - Forest Investigative Site, Anaheim, California
  - Forest Investigative Site, Burbank, California
  - Forest Investigative Site, Lakewood, California
  - Forest Investigative Site, National City, California
  - Forest Investigative Site, Riverside, California
  - Forest Investigative Site, Sacramento, California
  - Forest Investigative Site, San Diego, California
  - Forest Investigative Site, Santa Monica, California
  - Forest Investigative Site, Tustin, California
  - Forest Investigative Site, Walnut Creek, California
  - Forest Investigative Site, Westlake Village, California
  - Forest Investigative Site, Boulder, Colorado
  - Forest Investigative Site, New Britain, Connecticut
  - Forest Investigative Site, Bradenton, Florida
  - Forest Investigative Site, Brandon, Florida
  - Forest Investigative Site, DeLand, Florida
  - Forest Investigative Site, Hollywood, Florida
  - Forest Investigative Site, Jacksonville, Florida
  - Forest Investigative Site, Miami, Florida
  - Forest Investigative Site, Orlando, Florida
  - Forest Investigative Site, Pembroke Pines, Florida
  - Forest Investigative Site, Tampa, Florida
  - Forest Investigative Site, West Palm Beach, Florida
  - Forest Investigative Site, Honolulu, Hawaii
  - Forest Investigative Site, Boise, Idaho
  - Forest Investigative Site, Wichita, Kansas
  - Forest Investigative Site, Covington, Louisiana
  - Forest Investigative Site, Owings Mills, Maryland
  - Forest Investigative Site, St Louis, Missouri
  - Forest Investigative Site, West Caldwell, New Jersey
  - Forest Investigative Site, Albuquerque, New Mexico
  - Forest Investigative Site, New York, New York
  - Forest Investigative Site, Charlotte, North Carolina
  - Forest Investigative Site, Greenville, North Carolina
  - Forest Investigative Site, Winston-Salem, North Carolina
  - Forest Investigative Site, Cleveland, Ohio
  - Forest Investigative Site, Kettering, Ohio
  - Forest Investigative Site, Tulsa, Oklahoma
  - Forest Investigative Site, Duncansville, Pennsylvania
  - Forest Investigative Site, Philadelphia, Pennsylvania
  - Forest Investigative Site, Columbia, South Carolina
  - Forest Investigative Site, Memphis, Tennessee
  - Forest Investigative Site, Dallas, Texas
  - Forest Investigative Site, Lake Jackson, Texas
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Salt Lake City, Utah
  - Forest Investigative Site, Virginia Beach, Virginia
  - Forest Investigative Site, Tacoma, Washington